CLINICAL TRIAL: NCT06158815
Title: Investigation of the Effects of Proprioceptive Neuromuscular Facilitation Exercises on Fatigue, Muscle Strength and Functional Parameters in Patients With Myasthenia Gravis
Brief Title: Investigation of the Effects of Proprioceptive Neuromuscular Facilitation Exercises in Patients With Myasthenia Gravis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ridvan muhammed adin, Master of Science, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-22017
Record Dates: First submitted 2023-11-22; First posted 2023-12-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Participants in the control group will be placed on a waiting list without any intervention during the 6-week study period.
- exercise group (Experimental): Participants in the exercise group will have face-to-face Proprioceptive Neuromuscular Facilitation Exercises during the 6-week study period.
  Interventions: Other: proprioceptive neuromuscular facilitation exercise

INTERVENTIONS:
Other: proprioceptive neuromuscular facilitation exercise — The basic principle of Proprioceptive Neuromuscular Facilitation exercises, which is defined as facilitating the responses of the neuromuscular mechanism by stimulating the proprioceptors, is that the movements in the human body have a rotational and oblique character and that a greater response can be obtained with movement against maximum resistance. It is aimed to achieve improvement in strength and movement ability through hand contacts, visual and verbal stimuli.
  Arms: exercise group

SUMMARY:
The goal of this clinical trial is to investigate of the effects of proprioceptive neuromuscular facilitation exercises on fatigue, muscle strength and functional parameters in patient with Myasthenia Gravis. The main questions it aims to answer are:

* Do proprioceptive neuromuscular facilitation exercises reduce fatigue in patients with Myasthenia Gravis?
* Do proprioceptive neuromuscular facilitation exercises increase muscle strength in patients with Myasthenia Gravis?
* Do proprioceptive neuromuscular facilitation exercises improve functional parameters in patients with Myasthenia Gravis?
* How well can patients with Myasthenia Gravis tolerate proprioceptive neuromuscular facilitation exercises? Participants will be divided into 2 groups as control group and exercise group with block randomization method. In this single-blind randomized controlled study, the participants in the control group will be placed on a waiting list without any intervention during the 6-week study period and at the end of the study, the interventions applied to the exercise group will be applied exactly the same. Proprioceptive neuromuscular facilitation exercises will be applied to the exercise group 3 days a week, 1 hour a day for 6 weeks. Individuals will be evaluated at the beginning and at the end of the study.

Researchers will compare exercise and control group to see if there are effects of proprioceptive neuromuscular exercises patients with Myasthenia Gravis.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being between the ages of 18-65
* It must be confirmed by the Neurologist that the patient has been diagnosed with adult onset and Achr+ generalized Myasthenia Gravis and has been in a stable condition for the last 6 months.
* Being in class II or III according to the American Myasthenia Gravis Foundation Clinical Classification

Exclusion Criteria:

* Having a cognitive problem or having a Mini Mental Test score below 24
* Change in the type and dose of medical treatment within the last 6 months
* Having another cardiorespiratory, metabolic, systemic, rheumatological, orthopaedic and neurological disease (unstable and at a level that prevents participation in the exercise programme) in addition to Myasthenia Gravis
* Having a body mass index below 17 kg/m2 and above 30 kg/m2
* Having participated in any physiotherapy program any intervention study for the last 6 months
* Having undergone pregnancy, birth or surgical operation in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
chalder fatigue scale | baseline and immediately after the intervention
  It is an easy, fast and useful scale that evaluates fatigue through self-report. The final version of the scale consists of a total of 11 items, including a 7-item physical fatigue subsection and a 4-item mental fatigue subsection. The individual is asked to respond to the statements using a four-point Likert scale (less than usual, as much as usual, more than usual, much more than usual). Each item is scored between 0-3 and the total score varies between 0-33.
Fatigue Impact Scale | baseline and immediately after the intervention
  It is a multidimensional scale that evaluates the physical, cognitive and social effects of fatigue. The scale consists of a total of 40 questions: 10 questions for the physical effects subscale, 10 questions for the cognitive effects subscale, and 20 questions for the social effects subscale. Individuals fill out the scale by taking their last month into consideration. All questions are scored from "0" (no problem) to "4" (very big problem). Higher scores indicate increased degree of fatigue.
fatigue severity scale | baseline and immediately after the intervention
  It is a self-report scale consisting of 9 items that evaluates the degree of fatigue severity in the last week. For each item, the patient marks the most appropriate statement on a 7-point Likert scale ranging from 7=strongly agree to 1=strongly disagree. The scores obtained from each item are added up and the total value is divided by 9.
Surface electromyography | baseline and immediately after the intervention
  Surface electromyography measurements will be performed to measure the electrical signals coming from the muscles to determine the fatigue of the muscles. It has been shown in the literature that fatigue can be measured by power spectrum analysis in neuromuscular diseases. For this purpose, surface electromyography electrodes will be placed on the vastus lateralis muscle and the middle part of the deltoideus muscle and the participants will be asked to make maximum isometric contraction for 30 seconds. Electromyography signals will be analyzed and median frequencies between 0-5 seconds and 25-30 seconds will be determined and recorded. Wireless surface electromyography sensors and portable data acquisition system will be used to record and store measurements (Delsys (Delsys Inc. Natick, Massachusetts, USA)).
Six Minute Walk Test | baseline and immediately after the intervention
  It will be applied to evaluate functional capacity in accordance with the guidelines of the American Thoracic Society. In this test, the participant is walked down a 30-meter straight corridor. Participants are asked to walk for 6 minutes at the maximum speed they can walk during the test. The total distance walked is recorded. The distance walked per minute will also be recorded during this test. From these data, physical fatigue will be calculated according to the fatigue ambulatory index formula.

SECONDARY OUTCOMES:
muscle strength | baseline and immediately after the intervention
  The upper extremity, lower extremity and neck muscles of the participants will be evaluated using a digital hand dynamometer (Lafayette Manual Muscle Tester Model 01165, Lafayette Instrument Company, Lafayette, IN, USA). Muscle strength measurements will be evaluated by applying a breaking test to measure maximum muscle strength, with a digital hand dynamometer placed between the patient's evaluating area and the physiotherapist's hand, depending on the principles and positions of manual muscle testing. In the upper extremities; shoulder flexors, shoulder extensors, shoulder abductors, elbow flexors and extensors, in the lower extremities; hip flexors, hip extensors, hip abductors, knee flexors and extensors will be evaluated. In the cervical region, both flexor and extensor muscle groups will be evaluated and recorded. Three measurements will be made for all muscles and the average value will be recorded.
functional capacity | baseline and immediately after the intervention
  Two timed performance tests will be used: the 30-second sit-to-stand test and the stair-climbing test. In the 30-second sit-to-stand test, the participant is asked to sit on a standard chair for 30 seconds. The participant is asked to sit and stand as many times as possible throughout the session. The number of repetitions performed within a 30-second period will be recorded. In the stair climbing test, the participant will be asked to climb 10 standard steps as quickly as possible. The time it takes to climb 10 steps will be recorded in seconds. Both methods are used to determine functional capacity in patients with Myasthenia Gravis.
Myasthenia Gravis-Activities of Daily Living Scale | baseline and immediately after the intervention
  It is a self-report scale consisting of eight items. It is designed to evaluate the functional performance of daily living activities impaired due to Myasthenia Gravis. Two of the items in the scale consist of ocular, three bulbar, one respiratory, and two extremity-related activities. Each item is rated from 0 to 3, and the total score range is 0 to 24. High scores indicate low independence.
Myasthenia Gravis Quality of Life Scale | baseline and immediately after the intervention
  It is a self-report scale consisting of fifteen items. It is designed to evaluate the change in quality of life due to Myasthenia Gravis. Items in the scale are scored between 0 and 4, and the total score range is 0-60. The higher the score, the worse the patient's perceived quality of life.
Myasthenia Gravis Composite Scale | baseline and immediately after the intervention
  It is a scale developed to determine disease severity, applied and scored by healthcare professionals. Myasthenia Gravis Composite Scale scoring is created by combining parts of three scales. Ocular evaluation was obtained from the Quantitative Myasthenia Gravis Scale, bulbar and neck flexion evaluations were obtained from the Myasthenia Gravis Activity of Daily Living Scale, and muscle strength tests were obtained from the Manual Muscle Test scale. Total score varies between 0-50. Higher scores indicate increased disease severity.
visual analog scale | immediately after the intervention
  How well patients can tolerate Proprioceptive Neuromuscular Facilitation Exercises and their satisfaction with the treatment will be evaluated with 4 visual analog scales. Visual Analogue Scale consists of a 100 mm line. At each end of the line, there are two opposing statements about the situation to be evaluated. The participant is asked to mark the point on the visual analog scale line that best reflects his or her feelings. The point marked by the participant is measured in cm or mm from the end point with the help of a ruler.

CONTACTS AND LOCATIONS:
Overall Officials: sevim erdem özdamar, Professor, Principal Investigator — Hacettepe University; yeliz salcı, Assoc. Prof., Study Chair — Hacettepe University; rıdvan m adın, M.Sc., Study Chair — Hacettepe University; ayla fil balkan, Assoc. Prof., Study Chair — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No